CLINICAL TRIAL: NCT03001414
Title: Study of Angiogenic Cell Therapy for Progressive Pulmonary Hypertension: Intervention With Repeat Dosing of eNOS-enhanced EPCs
Brief Title: Study of Angiogenic Cell Therapy for Progressive Pulmonary Hypertension
Acronym: SAPPHIRE
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lower than anticipated enrollment
Sponsor: Northern Therapeutics (Industry)
Collaborators: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-PAH002
Record Dates: First submitted 2016-12-15; First posted 2016-12-23 (Estimated); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Hypertension,Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo followed by Autologous EPCs transfected with eNOS (Experimental): 4 monthly IV injections of Placebo (Plasma-Lyte A) during Course 1 followed by 4 monthly IV injections of Autologous EPCs transfected with human eNOS (total of 80 million cells) during Course 2
  Interventions: Biological: Placebo followed by Autologous EPCs transfected with human eNOS
- Autologous EPCs transfected with eNOS followed by Placebo (Experimental): 4 monthly IV injections of Autologous EPCs transfected with human eNOS (total of 80 million cells) during Course 1 followed by 4 monthly IV injections of Placebo (Plasma-Lyte A) during Course 2
  Interventions: Biological: Autologous EPCs transfected with human eNOS followed by Placebo
- Autologous EPCs transfected with eNOS (Experimental): 4 monthly IV injections of Autologous EPCs transfected with human eNOS in Course 1 followed by 4 monthly injections of Autologous EPCs transfected with human eNOS in Course 2 (total of 160 million cells)
  Interventions: Biological: Autologous EPCs transfected with human eNOS

INTERVENTIONS:
Biological: Placebo followed by Autologous EPCs transfected with human eNOS — 4 doses of placebo in first 6 months followed by 4 doses of autologous EPCs transfected with eNOS in second 6 months
  Arms: Placebo followed by Autologous EPCs transfected with eNOS
Biological: Autologous EPCs transfected with human eNOS followed by Placebo — 4 doses of autologous EPCs transfected with eNOS in first 6 months followed by 4 doses of placebo in second 6 months
  Arms: Autologous EPCs transfected with eNOS followed by Placebo
Biological: Autologous EPCs transfected with human eNOS — 4 doses of autologous EPCs transfected with eNOS in first 6 months which is repeated in second 6 months
  Arms: Autologous EPCs transfected with eNOS

SUMMARY:
The SAPPHIRE clinical trial seeks to establish the efficacy and safety of repeated monthly dosing of autologous EPCs transfected with human eNOS (heNOS) in patients with symptomatic severe PAH on available PAH-targeted medical therapy.

DETAILED DESCRIPTION:
SAPPHIRE will use autologous progenitor cell-based gene delivery to enhance lung microvascular repair and regeneration in patients with severe symptomatic PAH. A total of 45 patients will be enrolled in this multi-centre, late phase, randomized, double-blind, placebo-controlled, 3-arm protocol. Up to nine centres across Canada will participate.

Consented study participants who meet all eligibility criteria during the screening period will be scheduled to undergo apheresis. Following successful apheresis collection and receipt of the cell samples by the cell manufacturing facility, randomization will take place though a web-based system. Manufacturing of the cell therapy product will then be performed by the cell manufacturing facility according to the assigned treatment allocation:

Arm 1: Placebo (Plasma-Lyte A; 4 monthly IV infusions) in Course 1 (1st 6 months) followed by Autologous EPCs transfected with human eNOS in Course 2 (2nd 6 months; 4 monthly IV infusions)

Arm 2: Autologous EPCs transfected with human eNOS in Course 1 (1st 6 months; 4 monthly IV infusions) followed by Placebo (Plasma-Lyte A) in Course 2 (2nd 6 months; 4 monthly IV infusions)

Arm 3: Autologous EPCs transfected with human eNOS in Course 1 (1st 6 months; 4 monthly IV infusions) followed by a repeat dosing with Autologous EPCs transfected with human eNOS in Course 2 (2nd 6 months; 4 monthly IV infusions)

Approximately 5-9 days later, the study product will be transported to the investigative site where the initial treatment will be delivered to the study participant in an outpatient setting which is equipped for continuous monitoring of vital signs and oxygen saturation. Participants will subsequently be monitored for a minimum of 1 hour and discharged from the clinic once judged by the study investigator to be clinically stable.

Treatment and follow-up assessments will take place over a 12-month period (11 study visits in total). Once the 12-month trial data collection is completed, the trial will convert to a registry with the goal of collecting long-term safety information through annual telephone contacts for 10 years. Participants will be permitted to enroll in other clinical trials during the registry period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, ≤ 80 years
* Established diagnosis of PAH due to the following:

  * Idiopathic or heritable PAH;
  * Scleroderma associated PAH (limited or diffuse);
  * Drugs (anorexigens) or toxins;
  * Congenital heart defects (atrial septal defects, ventricular septal defects, and patent ductus arteriosus) repaired ≥ 1 years
* World Health Organization (WHO) functional class II, III, or IV on appropriate stable therapy for PAH for at least 3 months prior to the screening period and up until randomization, apart from modification of anticoagulant or diuretic dosages, or small adjustments in prostaglandin dose that are considered by the Investigator to be consistent with stable parenteral therapy.
* Able to walk unassisted (oxygen use allowed). Aids for carrying oxygen (such as a wheel chair or walker) are permitted provided they are not also required as mobility aids.
* An average 6-Minute Walk Distance (6MWD) of ≥ 125 meters and ≤ 440 meters on two consecutive tests during the Screening period
* Previous diagnostic right heart cardiac catheterization (RHC) at the time of PAH diagnosis with findings consistent with PAH: specifically, mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg (at rest); pulmonary vascular resistance (PVR) ≥ 3 WU; pulmonary capillary wedge pressure (PCWP) (or left ventricular end diastolic pressure) ≤12 mmHg if PVR ≥ 3 to < 5 Woods Units (WU), or pulmonary capillary wedge pressure (PCWP) (or left ventricular end diastolic pressure) ≤ 15 mmHg if PVR ≥ 5 WU. If repeat testing has occurred since initial diagnosis, the most recent results should be used.
* Echocardiography performed within 12 months prior to the Screening Period confirming a left atrial volume index (LAVI) of ≤ 34 ml/m2 and the absence of any clinically significant left heart disease including evidence of more than mild left-sided valvular heart disease, systolic or diastolic left ventricular dysfunction
* Ventilation and perfusion (VQ) nuclear scan performed as part of the initial workup to establish the diagnosis of PAH showing absence (i.e. low probability) of pulmonary embolism. If repeat testing has occurred since initial diagnosis, the most recent results should be used. In the absence of a VQ scan to establish eligibility, a CT angiogram that has been reviewed by a radiologist with expertise in the work up for pulmonary endarterectomy and deemed negative for chronic thromboembolic disease may be used instead.
* Pulmonary function tests conducted within 2 years prior to the Screening Period to confirm: total lung capacity (TLC) ≥ 65% the predicted value; and forced expiratory volume at one second (FEV1) of ≥ 65% the predicted value
* Must have a resting arterial oxygen saturation (SaO2) ≥88% with or without supplemental oxygen as measured by pulse oximetry at the Screening Visit
* Must not be enrolled in an exercise training program for pulmonary rehabilitation within 3 months prior to the Screening Visit and must agree not to enroll in an exercise training program for pulmonary rehabilitation during the Screening Period and the first 6 months of the study. Participants enrolled in an exercise program for pulmonary rehabilitation 3 months prior to screening may enter the study if they agree to maintain their current level of rehabilitation for the first 6 months of the study
* Women of child-bearing potential (defined as less than 1 year post-menopausal and not surgically sterile) must be practicing abstinence or using two highly effective methods of contraception (defined as a method of birth control that results in a low failure rate, i.e., less than 1% per year, such as approved hormonal contraceptives, barrier methods [such as a condom or diaphragm] used with a spermicide, or an intrauterine device). Subjects must have a negative ß-human chorionic gonadotropin (hCG) pregnancy test during the Screening period and negative urine pregnancy test results at all other study visits
* Must be willing and able to comply with study requirements and restrictions.

Exclusion Criteria:

* Pregnant or lactating
* PAH related to any condition not covered under inclusion criteria, including but not limited to pulmonary venous hypertension, pulmonary veno-occlusive disease, pulmonary capillary hemangiomatosis, or chronic thromboembolic pulmonary hypertension
* Evidence of more than mild interstitial lung disease on Chest CT within the last 5 years (last 3 years for patients with scleroderma associated PAH)
* Treatment with an investigational drug, device or therapy within 3 months prior to the screening period or is scheduled to receive an investigational drug, device or therapy during the course of the study
* Any musculoskeletal disease or any other disease that would significantly limit ambulation
* Unrepaired or recently repaired (< 1 year) congenital systemic-to-pulmonary shunt other than patent foramen ovale
* Patients having three or more of the following four AMBITION study heart failure preserved ejection fractio (HFpEF) risk factors will be excluded:

  * BMI ≥ 30 kg/m2,
  * History of essential hypertension,
  * Diabetes mellitus (any type)
  * Historical evidence of significant coronary artery disease (CAD) by any one of the following:

    * History of myocardial infarction (MI)
    * History of percutaneous coronary intervention (PCI)
    * Prior coronary angiography evidence of CAD (>50% stenosis in ≥1 vessel)
    * Previous positive Stress Test
    * Previousoronary artery bypass grafting (CABG)
    * Stable angina
* Creatinine clearance <30 ml/min (using the Cockroft-Gault formula) or requires hemodialysis
* Inability to undergo the apheresis procedure due to poor venous access or laboratory tests that are not within acceptable ranges (not including international normalized ratio (INR) for patients on Coumadin)
* Childs-Pugh class C liver cirrhosis
* Previous atrial septostomy
* Any other clinically significant illness or abnormal laboratory values (measured during the screening period) that, in the opinion of the Investigator, might put the subject at risk of harm during the study or might adversely affect the interpretation of the study data
* Anticipated survival less than 1 year due to concomitant disease
* History of cancer in the past 5 years (except for low grade and fully resolved non-melanoma skin cancer)
* Results during screening consistent with current infection with HIV, Hepatitis B (HBV) or C (HCV), human T-cell lymphotropic virus (HTLV- I/II) or syphilis
* Systemic arterial systolic blood pressure < 85 mm Hg
* Known allergy to gentamicin or amphotericin
* Patients who have participated in any gene therapy study or an angiogenic growth factor protein study
* Patients unable to provide informed consent and comply with the visit schedule.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duncan J Stewart, MD FRCPC, Study Director — Northern Therapeutics, Inc.
Locations (4):
- Canada (4):
  - Peter Lougheed Center, University of Calgary, Calgary, Alberta
  - London Health Sciences Center, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral from specialized Pulmonary Arterial Hypertension clinics at 6 participating study sites between October 2017 and August 2022. The first participant was enrolled on November 24, 2017 and the last participant was enrolled on August 24, 2022.
Pre-assignment Details: Of 22 enrolled participants, 12 met the required inclusion criteria and were randomized to receive treatment with the study product.
Groups:
- Arm 1 - Placebo Followed by Autologous Endothelial Progenitor Cells (EPCs) Transfected With eNOS: 4 monthly IV injections of Placebo (Plasma-Lyte A) during Course 1 followed by 4 monthly IV injections of Autologous EPCs transfected with human eNOS (total of 80 million cells) during Course 2
  Placebo followed by Autologous EPCs transfected with human eNOS: 4 doses of placebo in first 6 months followed by 4 doses of autologous EPCs transfected with eNOS in second 6 months
- Arm 2 - Autologous EPCs Transfected With Endothelial NO-synthase (eNOS) Followed by Placebo: 4 monthly IV injections of Autologous EPCs transfected with human eNOS (total of 80 million cells) during Course 1 followed by 4 monthly IV injections of Placebo (Plasma-Lyte A) during Course 2
  Autologous EPCs transfected with human eNOS followed by Placebo: 4 doses of autologous EPCs transfected with eNOS in first 6 months followed by 4 doses of placebo in second 6 months
- Arm 3 - Autologous EPCs Transfected With eNOS: 4 monthly IV injections of Autologous EPCs transfected with human eNOS in Course 1 followed by 4 monthly injections of Autologous EPCs transfected with human eNOS in Course 2 (total of 160 million cells)
  Autologous EPCs transfected with human eNOS: 4 doses of autologous EPCs transfected with eNOS in first 6 months which is repeated in second 6 months
Period: Overall Study
Arm/Group | Arm 1 - Placebo Followed by Autologous Endothelial Progenitor Cells (EPCs) Transfected With eNOS | Arm 2 - Autologous EPCs Transfected With Endothelial NO-synthase (eNOS) Followed by Placebo | Arm 3 - Autologous EPCs Transfected With eNOS
Started | 5 | 3 | 4
Completed | 5 | 3 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Followed by Autologous EPCs Transfected With eNOS | Autologous EPCs Transfected With eNOS Followed by Placebo | Autologous EPCs Transfected With eNOS | Total
Number analyzed (Participants) | 5 | 3 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (15.4) | 48.7 (5.8) | 55 (4.3) | 55.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 10
  Male | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 4 | 3 | 3 | 10
  Indigenous | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 0 | 1
Pulmonary arterial hypertension (PAH) Diagnosis [Count of Participants; unit: Participants]
  Idopathic/Hereditable | 3 | 2 | 2 | 7
  Drugs/Toxins | 2 | 0 | 1 | 3
  Congenital Heart Defects | 0 | 1 | 1 | 2
Oxygen Saturation [Mean (Standard Deviation); unit: Percent] | 93.4 (3.7) | 95.0 (3.0) | 95.0 (3.6) | 94.3 (3.3)
6 Minute Walk Test Distance [Mean (Standard Deviation); unit: Meters] | 345.4 (71.48) | 381.0 (11.53) | 329.25 (78.08) | 348.92 (60.57)
Concurrent Medications [Count of Participants; unit: Participants]
  PDE5 Inhibitor | 4 | 2 | 1 | 7
  Endothelin Receptor Antagonist | 3 | 3 | 4 | 10
  Soluble GC Stimulator | 1 | 1 | 0 | 2
  Prostaglandin Intravenous | 1 | 1 | 0 | 2
  Dual Therapy | 3 | 1 | 2 | 6
  Triple Therapy | 1 | 1 | 2 | 4
Comorbidities [Count of Participants; unit: Participants]
  Hypertension | 2 | 0 | 1 | 3
  Asthma | 2 | 1 | 0 | 3
  Emphysema | 1 | 0 | 0 | 1
  Obstructive Sleep Apnea | 0 | 0 | 1 | 1
  Gastrointestinal Reflux | 2 | 1 | 3 | 6
  Type 2 Diabetes | 1 | 0 | 0 | 1
  Hypothyroidism | 2 | 0 | 0 | 2
  Morbid Obesity | 0 | 0 | 1 | 1
  Seasonal Allergies | 1 | 0 | 0 | 1
Hemodynamic Parameters [Mean (Standard Deviation); unit: mmHg]
  Mean pulmonary arterial pressure (PAP) (mmHg) | 79 (13) | 74 (4) | 80 (15) | 78 (11)
  PCWP (mmHg) | 11 (6) | 9.7 (7.2) | 8.5 (4.8) | 9.9 (5.5)
Cardiac Output [Mean (Standard Deviation); unit: L/min] | 5.39 (1.36) | 4.55 (0.41) | 5.25 (2.26) | 5.13 (1.49)
Pulmonary vascular resistance (PVR) [Mean (Standard Deviation); unit: WU] | 6.18 (2.87) | 7.87 (2.87) | 7.95 (3.26) | 7.19 (2.78)

OUTCOME MEASURES:

1. Primary Outcome: Change in 6 Minute Walk Distance (6MWD) From Baseline
Description: Change was calculated as the distance walked at 6 months minus the distance at baseline.
Time Frame: Baseline, 6 months
Population: All participants for whom the 6MWD test was completed at baseline and 6 months.
Measure: Mean (Standard Deviation); unit: Meters
Groups:
- Arm 1 - Placebo During First 6 Months: 4 monthly IV injections of Placebo (Plasma-Lyte A) during Course 1
- Arm 2 and 3 During First 6 Months: 4 monthly IV injections with EPCs transfected with eNOS during Course 1
Arm/Group | Arm 1 - Placebo During First 6 Months | Arm 2 and 3 During First 6 Months
Number analyzed (Participants) | 5 | 7
Meters | 22.3 (38.49) | 36.00 (31.11)
Statistical Analysis 1: Comparison: Arm 1 - Placebo During First 6 Months vs Arm 2 and 3 During First 6 Months; Due to sample size restriction, the primary analysis plan was modified to analyze change from baseline to each time point using repeated measures of ANOVA; Test type: Superiority; p = 0.42, ANOVA; Global test of difference between the arms analyzed as absolute change from baseline; Mean Difference (Final Values) = 13.70, 95% CI 2-sided [-20.08 to 47.48], Standard Error of Mean 16.69
Statistical Analysis 2: Comparison: Arm 1 - Placebo During First 6 Months vs Arm 2 and 3 During First 6 Months; Calculation of raw change from baseline in meters using non-parametric Wilcoxon test; Test type: Superiority; p = 0.57, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 13.70
Statistical Analysis 3: Comparison: Arm 1 - Placebo During First 6 Months vs Arm 2 and 3 During First 6 Months; Test type: Superiority; p = 0.53, Wilcoxon (Mann-Whitney); Secondary analysis of primary outcome using non-parametric Wilcoxon test of percent change from baseline; Mean Difference (Final Values) = 4.55

2. Secondary Outcome: Change in 6 Minute Walk Distance (6MWD) From Baseline
Description: Comparison of change from baseline after delivery of 4 versus 8 doses of study product (Arms 2 versus Arm 3). Change was calculated by the distance walked at 12 months minus the distance walked at baseline.
Time Frame: Baseline and 12 months
Population: All participants in Arm 2 and 3 for whom the 6MWD test results were recorded at baseline and 12 months.
Measure: Mean (Standard Deviation); unit: Meters
Groups:
- Arm 2 - Autologous EPCs Transfected With eNOS Followed by Placebo: 4 monthly IV doses of autologous EPCs transfected during the first 6 months followed by 4 monthly IV doses of placebo during the second 6 months.
- Arm 3 - Autologous EPCs Transfected With eNOS: 8 monthly !V injections of autologous EPCs transfected with eNOS over 12 months
Arm/Group | Arm 2 - Autologous EPCs Transfected With eNOS Followed by Placebo | Arm 3 - Autologous EPCs Transfected With eNOS
Number analyzed (Participants) | 3 | 4
Meters | 49.3 (11.68) | 7.33 (9.02)
Statistical Analysis 1: Comparison: Arm 2 - Autologous EPCs Transfected With eNOS Followed by Placebo vs Arm 3 - Autologous EPCs Transfected With eNOS; Comparison of these arms is in accordance with the statistical analysis plan; Test type: Superiority — Change from baseline calculated in meters using non-parametric analysis; p = 0.10, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 41.97

3. Secondary Outcome: Change in 6 Minute Walk Distance (6MWD) From Baseline
Description: Comparison of change from baseline to assess durability of any measured improvement (Arm 2 only). Durability of any improvement at 3 versus 9 months post-treatment (measured at 6 and 12 months).
Time Frame: Baseline, 6 months, 12 months
Population: All participants in Arm 2 for whom the 6MWD test results were recorded at baseline, 6 months, and 12 months.
Measure: Mean (Standard Deviation); unit: Meters
Groups:
- 4 Monthly Doses of Autologous EPCs Transfected With eNOS Followed by 4 Monthly Doses of Placebo: 4 monthly IV doses of autologous EPCs transfected with eNOS during the first 6 months followed by 4 monthly IV doses of placebo during the second 6 months.
Arm/Group | 4 Monthly Doses of Autologous EPCs Transfected With eNOS Followed by 4 Monthly Doses of Placebo
Number analyzed (Participants) | 3
Meters
  Change from baseline to 6 months | 47.3 (32.50)
  Change from baseline to 12 months | 49.3 (11.68)
Statistical Analysis 1: Comparison: 4 Monthly Doses of Autologous EPCs Transfected With eNOS Followed by 4 Monthly Doses of Placebo; The selected arm for this outcome measure is in accordance with the statistical analysis plan; Test type: Superiority; p = 0.50, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 5.6

4. Secondary Outcome: Change in 6MWD From Baseline
Description: Incremental effect of 8 versus 4 doses at 6 and 12 months in arm 3 only.
Time Frame: Baseline, 6 months, 12 months
Population: Change was calculated as the distance at 6 months minus the distance at baseline and the distance at 12 months minus the distance at baseline
Measure: Mean (Standard Deviation); unit: Meters
Groups:
- Arm 3 -: 4 monthly IV injections of eNOS-transfected EPCs in 1st 6 months followed by a repeat of 4 monthly IV injections of eNOS-transfected EPCs in 2nd 6 months.
Arm/Group | Arm 3 -
Number analyzed (Participants) | 4
Meters
  Change from baseline to 6 months | 30.25 (33.61)
  Change from baseline to 12 months | 7.33 (9.02)
Statistical Analysis 1: Comparison: Arm 3 -; Selection of the arm for analysis of this outcome measure is in accordance with the statistical analysis plan; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney); Comparison of change from baseline in meters at 6 and 12 months; Mean Difference (Final Values) = 22.92

5. Secondary Outcome: Change in Pulmonary Vascular Resistance From Baseline
Description: Comparison of change from baseline after 4 doses of study product (Arms 2 and 3 versus Arm 1)
Time Frame: 6 months
Population: Participants in Arm 1 and Arm 2 and 3 combined for whom PVR was measured at baseline and 6 months.
Measure: Mean (Standard Deviation); unit: Wood Units (WU)
Groups:
- Arm 2 and 3 - eNOS-transfected Cells During First 6 Months: 4 monthly IV injections with EPCs transfected with eNOS during course 1
Arm/Group | Arm 1 - Placebo During First 6 Months | Arm 2 and 3 - eNOS-transfected Cells During First 6 Months
Number analyzed (Participants) | 5 | 7
Wood Units (WU) | 0.444 (1.18) | 0.576 (2.07)
Statistical Analysis 1: Comparison: Arm 1 - Placebo During First 6 Months vs Arm 2 and 3 - eNOS-transfected Cells During First 6 Months; Selection of the arms for analysis of this outcome measure is in accordance with the statistical analysis plan; Test type: Superiority; p = 0.81, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.132

6. Secondary Outcome: Change in Pulmonary Vascular Resistance From Baseline
Description: Comparison of change from baseline after delivery of 4 versus 8 doses of study product (Arm 2 versus Arm 3)
Time Frame: Baseline and 12 months
Population: Participants in Arm 2 and Arm 3 for whom the PVR was measured at baseline and 12 months
Measure: Mean (Standard Deviation); unit: Wood Units (WU)
Groups:
- Arm 2 - eNOS-transfected EPCs During First 6 Months: 4 monthly IV injections of Placebo (Plasma-Lyte A) during Course 1
- Arm 3 - eNOS-transfected Cells During First and Second 6 Months: 4 monthly IV injections with EPCs transfected with eNOS during course 1 and course 2
Arm/Group | Arm 2 - eNOS-transfected EPCs During First 6 Months | Arm 3 - eNOS-transfected Cells During First and Second 6 Months
Number analyzed (Participants) | 3 | 4
Wood Units (WU) | 0.09 (1.81) | 2.15 (3.09)
Statistical Analysis 1: Comparison: Arm 2 - eNOS-transfected EPCs During First 6 Months vs Arm 3 - eNOS-transfected Cells During First and Second 6 Months; Selection of the arms for analysis of this outcome measure is in accordance with the statistical analysis plan; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2.06

7. Secondary Outcome: Incremental Effect of 8 Versus 4 Doses of Cell Therapy Product on PVR
Description: Incremental effect of 8 versus 4 doses of cell therapy product on PVR at 6 and 12 months (Arm 3 only)
Time Frame: 6 and12 months
Population: All participants in whom the PVR was measurement at baseline, 6, and 12 months.
Measure: Mean (Standard Deviation); unit: Wood Units (WU)
Groups:
- Arm 3 - eNOS-transfected Cells in 1st and 2nd 6 Months: 4 monthly IV injections of eNOS-transfected EPCs in 1st 6 months followed by a repeat of 4 monthly IV injections of eNOS-transfected EPCs in 2nd 6 months.
Arm/Group | Arm 3 - eNOS-transfected Cells in 1st and 2nd 6 Months
Number analyzed (Participants) | 4
Wood Units (WU)
  Baseline to 6 months | 0.76 (0.87)
  Baseline to 12 months | 2.15 (3.09)
Statistical Analysis 1: Comparison: Arm 3 - eNOS-transfected Cells in 1st and 2nd 6 Months; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.39

8. Secondary Outcome: Change in Quality of Life Measures From Baseline
Description: Comparison of change from baseline measured by the Short Form 36 (SF-36) Health Survey after delivery of 4 doses of study product (Arms 2 and 3 versus Arm 1).
  Scale used ranging from 0-100. Lower scores indicate more significant limitations.
Time Frame: Baseline and 6 months
Population: All participants in Arm 1 and Arms 2 and 3 combined for whom results of the SF-36 questionnaire were collected baseline and 6 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Arm 2 and 3 During First 6 Months: 4 monthly IV injections with EPCs transfected with eNOS
Arm/Group | Arm 1 - Placebo During First 6 Months | Arm 2 and 3 During First 6 Months
Number analyzed (Participants) | 5 | 7
score on a scale
  Physical Component | 2.78 (5.11) | 3.2 (10.71)
  Mental Component | -2.60 (11.32) | -2.50 (6.93)
Statistical Analysis 1: Comparison: Arm 1 - Placebo During First 6 Months vs Arm 2 and 3 During First 6 Months; Selection of the arms for analysis of this outcome measure is in accordance with the statistical analysis plan; Test type: Superiority; p = 1.0, Wilcoxon (Mann-Whitney); This analysis represents the results for the Physical Component score of the questionnaire; Mean Difference (Final Values) = 5.6
Statistical Analysis 2: Comparison: Arm 1 - Placebo During First 6 Months vs Arm 2 and 3 During First 6 Months; Selection of the arms for analysis of this outcome measure is in accordance with the statistical analysis plan; Test type: Superiority; p = 0.64, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.10 — This analysis represents the difference in score for the mental component of the questionnaire

9. Secondary Outcome: Change in Quality of Life Measures From Baseline
Description: Comparison in change from baseline measured by SF-36 Survey after delivery of 4 versus 8 doses of study product (Arm 2 versus Arm 3).
  Scale used ranging from 0-100. Lower scores indicate more significant limitations.
Time Frame: 12 months
Population: All participants in Arm 2 and 3 for whom results of the SF-36 questionnaire were collected baseline and 12 months.
Measure: Mean (Standard Deviation); unit: Change in Score
Arm/Group | Arm 2 - Autologous EPCs Transfected With eNOS Followed by Placebo | Arm 3 - Autologous EPCs Transfected With eNOS
Number analyzed (Participants) | 3 | 4
Change in Score
  Physical Component | 10.5 (2.78) | 2.5 (13.86)
  Mental Component | 14.3 (21.58) | -1.10 (9.10)
Statistical Analysis 1: Comparison: Arm 2 - Autologous EPCs Transfected With eNOS Followed by Placebo vs Arm 3 - Autologous EPCs Transfected With eNOS; Selection of the arms for analysis of this outcome measure is in accordance with the statistical analysis plan; Test type: Superiority; p = 0.40, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 8.0 — This analysis represents the difference in score for the physical component of the questionnaire
Statistical Analysis 2: Comparison: Arm 2 - Autologous EPCs Transfected With eNOS Followed by Placebo vs Arm 3 - Autologous EPCs Transfected With eNOS; Test type: Superiority; p = 0.23, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 15.4; This analysis represents the change in score for the mental component of the questionnaire

ADVERSE EVENTS:
Time Frame: Adverse event data collection took place during the 12-month treatment phase of the trial.
Arm/Group | Placebo Followed by Autologous EPCs Transfected With eNOS | Autologous EPCs Transfected With eNOS Followed by Placebo | Autologous EPCs Transfected With eNOS
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/3 | 1/4
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Followed by Autologous EPCs Transfected With eNOS (N=5) | Autologous EPCs Transfected With eNOS Followed by Placebo (N=3) | Autologous EPCs Transfected With eNOS (N=4)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) — Chest x-ray in ER confirmed pneumonia. Started on antibiotics and admitted for monitoring. Patient discharged with no further issues. This event was deemed not related to the study product by the Principal Investigator.
Volume Overload (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Diagnosed by right heart catheterization. Deemed not related to study product by Principal Investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Followed by Autologous EPCs Transfected With eNOS (N=5) | Autologous EPCs Transfected With eNOS Followed by Placebo (N=3) | Autologous EPCs Transfected With eNOS (N=4)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Swollen Left Eye Lid (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2) | 2 (5)
Severe Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Tonsil Exudate (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Loss of Balance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrophic Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Erosive Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Nose Bleed (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Sinusitis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Left Ankle Sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Allergy Symptoms (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Elevated Jugular Venous Pulse (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pulsatile Right Upper Quadrant Abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Right Ankle Edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Right Eye Stye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid Infection (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Increased Pulmonary Vascular Resistance (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Emesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Increased Frequency of Headaches (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (2)
Elevated C-Reactive Protein (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Warm feeling (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Weakness/Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Volume Overload (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Right Submandibular Firm Node (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Left Knee Meniscus Deterioration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the corona virus disease (COVID)-19 pandemic, the trial was stopped after only 12 of the planned 45 patients were enrolled and randomized. This resulted in insufficient power for a reliable statistical analysis and necessitated a change to the analysis methods.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication or presentation or results is to be made by the study sponsor within 18 months of trial completion. For publications or results communications after that time, Principal Investigators must provide a copy of the proposed manuscript or presentation to the study sponsor for review at least 45 days prior to submission for consideration of publication, and the sponsor may request removal of confidential information which is protected as intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03001414/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT03001414/SAP_001.pdf